CLINICAL TRIAL: NCT04260789
Title: Safety and Performance Evaluation of Seraph 100 Microbind Affinity Blood Filter (Seraph 100) in the Reduction of Pathogen Load From the Blood in Septic Patients With Suspected, Life-threatening Bloodstream Infection
Brief Title: Reduction of Pathogen Load From the Blood in Septic Patients With Suspected, Life-threatening Bloodstream Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ExThera Medical Europe BV (Industry)
Collaborators: ExThera Medical Corporation (Industry); Vivantes Clinic Neukölln (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP015
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Bloodstream Infection
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Intervention Model Description: Open randomized post-market trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Other): Treatment with Seraph Filter
  Interventions: Device: Seraph 100,The Microbind Affinity Blood Filter
- Control (No Intervention)

INTERVENTIONS:
Device: Seraph 100,The Microbind Affinity Blood Filter — Treatment with Seraph 100 in one arm
  Arms: Treatment

SUMMARY:
Safety and Performance Evaluation of Seraph 100 Microbind Affinity Blood Filter (Seraph 100) in the reduction of pathogen load from the blood in septic patients with suspected, life-threatening bloodstream infection

DETAILED DESCRIPTION:
With the lack of effective antibiotics for many bloodstream infections, and limited new anti-infectives in development, there is a significant unmet need for new approaches that can help treat drug-resistant infections, especially in patients at high risk. There is an unmet need for a safe and broad-spectrum hemoperfusion therapy that can quickly reduce bacterial load and shorten the duration of bacteremia, preferably without the need to first identifying the type of bacteria present in the blood. There is an emerging need to increase the efficacy of effective antibiotics, e.g., by using hemadsorption as adjunctive therapy, to by quickly reducing bacterial load while scavenging toxins released from bacteria. Finally, there is a medical growing need for an alternative therapy when no effective antibiotic is available.

Seraph 100 Microbind Affinity Blood Filter is used to reduce pathogen load during bloodstream infection. Bacteremia or bloodstream infection, also called BSI, occurs when a bacterial infection elsewhere in the body enters the bloodstream. This clinical condition can quickly become life-threatening and progress to sepsis. Sepsis is defined as life-threatening organ dysfunction caused by a dysregulated host response to infection (Singer et al., 2016).When sepsis occurs with extremely low blood pressure, it's called septic shock. Septic shock is fatal in many cases.

Sepsis can be triggered by many types of bacteremia although the exact source of the infection often cannot be determined. Some of the most common infections that lead to BSI are lung infections (i.e. pneumonia) and infections in the abdominal area. Patients who are already in the hospital for something else, such as a surgery, are at a higher risk of developing BSI. These infections are even more dangerous when the bacteria are already resistant to antibiotics. The National Institutes of Health (NIH) estimates that over 1 million Americans get sepsis each year. Between 28 and 50 percent of these patients may die from the condition.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with sepsis and suspected bloodstream infection
2. Be ≥ 18 years old and ≤ 90 years old
3. Adults receiving IV antibiotic therapy
4. Increase of at least two points of the Sequential Organ Failure Assessment (SOFA) score
5. Subjects that presents Procalcitonin (PCT) levels > 0,5 ng/mL

Exclusion Criteria:

1. Subject is currently participating in another clinical investigation
2. Pregnant or nursing subjects and those who plan pregnancy during the clinical investigation follow-up period
3. Presence of comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results
4. The first dose of the current antibiotic therapy was > 24 h before screening
5. Have Child-Pugh Class C cirrhosis
6. Have platelet count < 30.000/uL
7. Contraindications for heparin sodium for injection
8. Subjects demonstrating any contraindication for this treatment as described in the IFU

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2020-08-19 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of pathogens load | 4,5 hours +/- 30 min
  Reduction of pathogens load from the bloodstream during treatment

SECONDARY OUTCOMES:
All-cause mortality | 90 days
  All-cause mortality
Persistence/Recurrence of bacteremia | Day 1, day 2, day 7
  Measure persistence recurrence of bacteremia
Persistence/Recurrence of sepsis | Daily during ICU stay or at least day 1, day 2, day 7
  Measure persistence recurrence of sepsis
Organ dysfunction-free days | Daily during ICU stay or at least day 1, day 2, day 7
  Measure organ dysfunction free days
Change of Intensive Care Unit (ICU) complications | Daily during ICU stay or at least day 1, day 2, day 7
  Reduction of ICU complications
Ventilator-free days (VFDs) | Daily during ICU stay or at least day 1, day 2, day 7
  VFD
Length of stay (LOS) at ICU and hospital ward | During ICU and hospital ward stay or at least day 1, day 2, day 7
  Measure LOS

OTHER OUTCOMES:
Treatment emergent adverse events | Occurrence within the 90 days follow-up period
  N (%) of patients with treatment emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Herwig Gerlach, Prof., Principal Investigator — Vivantes Clinic Neukölln
Locations (25):
- Medical University of Innsbruck, Innsbruck, Austria
- Belgium (2):
  - Middelheim Hospital, Antwerp
  - Hôpital Erasme, Brussels
- France (3):
  - CHU Bocage Central, Dijon
  - Hospices Civils de Lyon, Lyon
  - Nouvel Hopital Civil, Strasbourg
- Germany (10):
  - Klinikum Aschaffenburg-Alzenau, Aschaffenburg
  - Vivantes Klinikum Neukölln, Berlin
  - Städtisches Klinikum Braunschweig GmbH, Braunschweig
  - Universität Witten-Herdecke, Cologne
  - Universitätsklinikum Essen (AöR), Essen
  - University Hospital Frankfurt, Frankfurt
  - Universitätsmedizin Greifswald, Greifswald
  - Asklepios Hospital St. Georg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universität Rostock, Rostock
- Italy (3):
  - Azienda Usl Toscana Centro, Florence
  - University Hospital, Pisa, Pisa
  - A.Gemelli University Hospital, Roma
- Netherlands (2):
  - Ziekenhuis Gelderse Vallei, Ede
  - Medisch Spectrum Twente, Enschede
- Jagiellonia University, Krakow, Poland
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinico San Carlos, Madrid
- Royal Surrey NHS Foundation Trust, London, United Kingdom